CLINICAL TRIAL: NCT00971087
Title: A Multicenter, Controlled Clinical Trial to Evaluate the Hologic Tomosynthesis Mammography
Brief Title: Multicenter Hologic Tomosynthesis Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hologic, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 09-03
Record Dates: First submitted 2009-09-02; First posted 2009-09-03 (Estimated); Results first posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
Keywords: Breast cancer; breast cancer screening
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subjects undergoing breast cancer screening (Other): The study population included both women undergoing routing annual mammography imaging and women undergoing a previously scheduled breast biopsy
  Interventions: Device: Hologic Selenia Dimensions Digital Breast Tomosynthesis System

INTERVENTIONS:
Device: Hologic Selenia Dimensions Digital Breast Tomosynthesis System — Subjects are exposed to the same number of investigational images collected on the investigational device (Selenia Dimensions Full Field Digital Mammography System). Subject enrollment occurs at the time subjects are being imaged for their standard of care mammographic work up (either screening mammogram or scheduled biopsy). All subjects undergoing a biopsy procedure will be imaged on the investigational device prior to their procedure.
  Other Names: Tomosynthesis; Tomo; Breast tomosynthesis; 3D Breast imaging; Selenia Dimensions; 2D plus 3D breast imaging

SUMMARY:
The purpose of this image acquisition study is to compare, in a Reader Study, the performance of Tomosynthesis (3D) to (2D FFDM) conventional images in an enriched retrospective reader study. Synthetic 2D images, generated from the tomosynthesis image, will be available to the readers to provide an over view of the anatomy similar to a scout view in CT imaging and to determine whether the 3-D images with the synthesized 2D overview are non-inferior to the 2-D images alone as determined by receiver operating characteristic (ROC) area under the curve.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Any ethnic origin
* No contraindication of routine bilateral mammography

Exclusion Criteria:

* Any contraindications to mammographic screening, including but not limited to:
* Significant existing breast trauma
* Pregnancy
* Lactating
* Previous surgical biopsy
* Previous breast cancer
* Placement of an internal breast marker
* Breast implants
* Unable to understand and execute written informed consent
* Breasts are too large to be imaged on the 24 cm by 29 cm detector with a single exposure

Ages: 18 Years to 110 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3521 (Actual)
Dates: Start 2009-09; Primary Completion 2011-09 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - Scottsdale Medical Imaging Ltd. (SMIL), Scottsdale, Arizona
  - Hoag Memorial Hospital, Newport Beach, California
  - UC Davis, Sacramento, California
  - Invision/Sally Jobe, Greenwood Village, Colorado
  - Boca Raton Community Hospital, Boca Raton, Florida
  - Memorial Florida, Hollywood, Florida
  - Luthern General - Advocate Health Care, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Spectrum Health, Grand Rapids, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Barnes Jewish, St Louis, Missouri
  - Elizabeth Wende Breast Clinic, Rochester, New York
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Magee Women's Hospital, Pittsburgh, Pennsylvania
  - York - Women's Imaging at Apple Hill, York, Pennsylvania
  - UTSW Center for Breast Care, Dallas, Texas
  - Memorial Hermann/ Memorial City, Houston, Texas
  - Intermountain Medical Imaging, Murray, Utah
  - Fletcher Allen Health Care, Burlington, Vermont
  - University of Virginia, Charlottesville, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects Undergoing Breast Cancer Screening: The study population included both women undergoing routing annual mammography imaging and women undergoing a previously scheduled breast biopsy.
  Subjects are exposed to the same number of investigational images collected on the investigational device (Selenia Dimensions Full Field Digital Mammography System). Subject enrollment occurs at the time subjects are being imaged for their standard of care mammographic work up (either screening mammogram or scheduled biopsy). All subjects undergoing a biopsy procedure will be imaged on the investigational device prior to their procedure
Period: Overall Study
Arm/Group | Subjects Undergoing Breast Cancer Screening
Started | 3521
Completed | 3521
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The population for this study was women undergoing breast cancer screening including those undergoing a screen mammogram or scheduled for a biopsy procedure.
  The arms/groups are combined for analysis- as analysis as centered on women undergoing breast cancer screening in general and not the clinical path which made the women eligible for the study.
Arm/Group | Subjects Undergoing Breast Cancer Screening
Number analyzed (Participants) | 3521
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3000
  >=65 years | 521
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3521
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 3521

OUTCOME MEASURES:

1. Primary Outcome: To Demonstrate Non-inferior ROC Performance as Measured by the Area Under the Curve When Comparing 3-Ds Plus 3-D Images to the 2-D Images.
Description: ROC performance as measured by the area under the curve when comparing 3-Ds plus 3-D images to the 2-D images.
Time Frame: At time of exam
Measure: Mean (Full Range); unit: Proportion
Groups:
- 3D + s2D: Investigational Image Set: Three Dimensional breast tomosynthesis images with a synthesized 2D image (3D + s2D)
- 2D FFDM: Two Dimensional full-field digital mammography (2D FFDM)
Arm/Group | 3D + s2D | 2D FFDM
Number analyzed (Participants) | 302 | 302
Proportion | 0.907 [0.887 to 0.925] | 0.867 [0.810 to 0.899]
Statistical Analysis 1: Comparison: 3D + s2D vs 2D FFDM; A multi-reader, multi-case ROC analysis will be used to compare 3D + s2D to 2D FFDM. The areas under the curve (AUC) will be used to compare ROC performance; Test type: Non-Inferiority or Equivalence — 3D + s2D will be considered non-inferior to 2D FFDM if the lower limit one-sided 95% CI for the difference in AUCs (3DS minus 2D FFDM) is greater than -0.05. That is, our null hypothesis is that the AUC for 3D + s2D is 0.05 less than the AUC for 2D FFDM. A difference of 0.05 is considered a clinically significant difference; p = 0.009, MRMC ROC Analysis

2. Secondary Outcome: Analysis of ROC Performance in Subjects With Dense Breasts
Description: The radiologist's POM case based score will be used to generate the 2D FFDM and 3DS ROC curves for women with dense breasts (defined as BIRADS density score of 3 or 4).
  Endpoint Analysis - A multi-reader, multi-case ROC analysis will be used to compare 3DS to 2D FFDM. The areas under the curve (AUC) will be used to compare ROC performance. 3DS will be considered non-inferior to 2D FFDM if the lower limit one-sided 95% CI for the difference in AUCs (3DS minus 2D FFDM) is greater than -0.05. A difference of 0.05 is considered a clinically significant difference.
Time Frame: At time of exam
Measure: Mean (Full Range); unit: Proportion
Groups:
- 3D + s2D: Investigational Image Set: Three Dimensional breast tomosynthesis images with synthesized 2D image (3D + s2D)
Arm/Group | 3D + s2D | 2D FFDM
Number analyzed (Participants) | 148 | 148
Proportion | 0.893 [0.859 to 0.929] | 0.848 [0.803 to 0.901]
Statistical Analysis 1: Comparison: 3D + s2D vs 2D FFDM; Test type: Non-Inferiority — A multi-reader, multi-case ROC analysis will be used to compare 3DS to 2D FFDM. The areas under the curve (AUC) will be used to compare ROC performance. 3DS will be considered non-inferior to 2D FFDM if the lower limit onesided 95% CI for the difference in AUCs (3DS minus 2D FFDM) is greater than -0.05; p = 0.045, MRMC ROC Analysis

3. Secondary Outcome: Analysis of Non-Cancer Recall Rate: 3DS Compared to 2D FFDM
Description: The non-cancer recall rate was measured for 3DS and 2D FFDM
Time Frame: at time of exam
Measure: Number; unit: percentage of recalls
Arm/Group | 3D + s2D | 2D FFDM
Number analyzed (Participants) | 76 | 76
percentage of recalls | 54.6 | 67.2

ADVERSE EVENTS:
Groups:
- Subjects Undergoing Breast Cancer Screening: The population for this study was women undergoing breast cancer screening including those undergoing a screen mammogram or scheduled for a biopsy procedure.
  The arms/groups are combined for reporting- centered on women undergoing breast cancer screening in general and not the clinical path which made the women eligible for the study.
Arm/Group | Subjects Undergoing Breast Cancer Screening
Serious Adverse Events (participants affected / at risk) | 0/3521
Other Adverse Events (participants affected / at risk) | 0/3521

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less